CLINICAL TRIAL: NCT05717387
Title: Effects of Intermittent Eating on Glucose Homeostasis in Prediabetes: A Randomized Clinical Trial
Brief Title: Intermittent Eating on Glucose Homeostasis in Prediabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Huijie Zhang, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2023-017
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: PreDiabetes; Obesity
Keywords: TRE; The 5:2 diet; Glucose Homeostasis; prediabetes; obesity
MeSH Terms: conditions — Prediabetic State; Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Time-restricted eating (Experimental): Participants in the TRE group will be instructed to eat during a window of 8 h/d (8 am to 4 pm)
  Interventions: Behavioral: Time-restricted eating
- the 5:2 diet (Experimental): Participants in the 5:2 diet group will be instructed to consume 500-600 kcal/d on fast days and eat ad libitum on feast days.
  Interventions: Behavioral: The 5:2 diet
- Control (No Intervention): Participants in the control group will receive a general lifestyle counseling.

INTERVENTIONS:
Behavioral: Time-restricted eating — Participants in the TRE group will be instructed to eat during a window of 8 h/d (8 am to 4 pm).
  Arms: Time-restricted eating
Behavioral: The 5:2 diet — Participants will be instructed to consume 500-600 kcal/d on fast days and eat ad libitum on feast days.
  Arms: the 5:2 diet

SUMMARY:
Prediabetes is a high-risk state for diabetes development, lifestyle modification is the cornerstone of diabetes prevention. Two novel types of intermittent fasting recently have received more attention: the 5:2 diet and time-restricted eating (TRE). TRE requires individuals to eat in a specified number of hours per day (typically 4 to 10 hours) without energy intake restriction. The 5:2 diet involves 5 feast days and 2 fast days per week; participants eat ad libitum without restriction on feast days while 25% of energy needs (approximately 500-800 kcal per day) are consumed on fast day. This randomized controlled trial aimed to evaluate the effect of TRE and the 5:2 diet on glucose homeostasis and cardiometabolic risk factors in prediabetes over 6 months compared to usual health care.

DETAILED DESCRIPTION:
Prediabetes is a high-risk state for diabetes development, lifestyle modification is the cornerstone of diabetes prevention. Two novel types of intermittent fasting recently have received more attention: the 5:2 diet and time-restricted eating (TRE). TRE requires individuals to eat in a specified number of hours per day (typically 4 to 10 hours) without energy intake restriction. The 5:2 diet involves 5 feast days and 2 fast days per week; participants eat ad libitum without restriction on feast days while 25% of energy needs (approximately 500-800 kcal per day) are consumed on fast day. Preliminary evidence suggests that both TRE and the 5:2 diet have beneficial effects on glucose control in type 2 diabetes. No much is known about the effects and molecular mechanisms by TRE or the 5:2 diet improves glucose homeostasis in prediabetes. This randomized controlled trial aimed to evaluate the effect of TRE and the 5:2 diet on glucose homeostasis and cardiometabolic risk factors in prediabetes over 6 months compared to usual health care. All eligible participants will participate in an 8-week run-in phase in which they are fed the low-calorie-diet. Participants who pass the run-in phase will be randomly assigned 1:1:1 to one of the three study groups (TRE, the 5:2 diet and control groups). Participants in the TRE group will be instructed to eat during a window of 8 h/d (8 am to 4 pm) over 12 months. Participants in the 5:2 diet group will be instructed to consume 500-600 kcal/d on fast days and eat ad libitum on feast days. Participants in the control group were instructed to receive usual health care.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18-75 years;
2. Prediabetes;
3. Body mass index (BMI)of 28.0 to 45.0 kg/m2;

Exclusion Criteria:

1. History of HIV, hepatitis B or C (self-report) or active pulmonary tuberculosis;
2. Diagnosis of type 1 and type 2 diabetes;
3. History of malignant tumors;
4. Serious liver dysfunction or chronic kidney disease (AST or ALT > 3 times the upper limit of normal, or eGFR<30 ml/min/1.73 m2);
5. History of serious cardiovascular or cerebrovascular disease (angina, myocardial infarction or stroke) in the past 6 months;
6. History of severe gastrointestinal diseases or gastrointestinal surgery in the past 12 months;
7. History of Cushing's syndrome, hypothyroidism, acromegaly, hypothalamic obesity;
8. Being a smoker or having been a smoker in the 3 months prior to their screening visit;
9. Taking medications affecting weight or energy intake/energy expenditure in the last 6 months, including weight loss medications, antipsychotic drugs or other medications as determined by the study physician;
10. Currently participating in weight loss programs;
11. Women who are pregnant or plan to become pregnant;
12. Patients who cannot be followed for 24 months (due to a health situation or migration);
13. Patients who are unwilling or unable to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in percent of time in range (glucose between 3.9-7.8mmol/L) over 6 months measured with continuous glucose monitoring. | Baseline to months 6

SECONDARY OUTCOMES:
Change in mean glucose levels | Baseline and months 6
Change in glycemic variability | Baseline and months 6
Change in percent of time below range | Baseline and months 6
  <3.9 mmol/L
Change in percent of time above range | Baseline and months 6
  >7.8 mmol/L
Change in resting metabolic rate | Baseline and months 6
  Resting metabolic rate will be assessed by indirect calorimetry.
Change in gut microbiome composition | Baseline and months 6
Change in bile acid level | Baseline and months 6
Change in body weight | Baseline and months 6
Change in body composition | Baseline and months 6
  Body composition will be assessed by DEXA.
Change in waist circumference | Baseline and months 6
Change in body mass index | Baseline and months 6
Change in liver fat | Baseline and months 6
  Liver fat will be assessed by liver Fibroscan.
Change in visceral fat | Baseline and months 6
  Visceral fat will be assessed by abdominal CT scan.
Change in Systolic Blood pressure | Baseline and months 6
Change in Diastolic Blood pressure | Baseline and months 6
Change in blood lipids | Baseline and months 6
Change in HbA1c | Baseline and months 6
Change in insulin sensitivity | Baseline and months 6
Change in β cell function | Baseline and months 6
Change in pulse wave velocity (PWV) | Baseline and months 6
Change in quality of life | Baseline and months 6
  Quality of life measured by the 12-item Short-Form Health Survey Questionnaire (SF-12)

CONTACTS AND LOCATIONS:
Overall Officials: Huijie Zhang, MD.PhD, Principal Investigator — Department of Endocrinology and Metabolism, Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China